CLINICAL TRIAL: NCT04886713
Title: Adipose Tissue Inflammation in the Development, Maintenance and Functional Impairments in Heart Failure With Preserved Ejection Fraction
Brief Title: Adipose Tissue Inflammation in HFpEF
Acronym: SLIM-HFpEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Clinical Investigator, Professor, Managing Senior Physician, Heart Center Leipzig - University Hospital
Other Study IDs: SLIM-HFpEF V1.0
Record Dates: First submitted 2021-03-25; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese HFpEF: Left ventricular-EF ≥ 50%, N-terminal-pro-brain natriuretic peptide (NT-proBNP) ≥ 125ng/l, evidence of structural heart diseases (diastolic dysfunction, Left ventricular-hypertrophy or Left atrial-dilatation) BMI ≥30 kg/m²
  Interventions: Diagnostic Test: Adipose and myocardial tissue sampling; Diagnostic Test: Cardiac magnetic resonance imaging; Diagnostic Test: Cardiopulmonary exercise testing
- Obese controls: No history of heart failure, Left ventricular-EF > 50% and NT-pro-BNP <125ng/l, BMI ≥ 30kg/m²
  Interventions: Diagnostic Test: Adipose and myocardial tissue sampling; Diagnostic Test: Cardiac magnetic resonance imaging; Diagnostic Test: Cardiopulmonary exercise testing
- Lean control: No history of heart failure, Left ventricular-EF > 50% and NT-pro-BNP <125ng/l, BMI < 30kg/m²
  Interventions: Diagnostic Test: Adipose and myocardial tissue sampling; Diagnostic Test: Cardiac magnetic resonance imaging; Diagnostic Test: Cardiopulmonary exercise testing

INTERVENTIONS:
Diagnostic Test: Adipose and myocardial tissue sampling — After median sternotomy tissue samples will be collected from the epicardial space, the abdominal wall and the myocardium.
Diagnostic Test: Cardiac magnetic resonance imaging — Magnetic resonance imaging will be performed at 1.5 Tesla ('Intera', Philips Medical Systems, Best, The Netherlands). All subjects will be examined in the supine position with initial anatomy scans to cover the thorax to the first sacral vertebrae. The magnetic resonance imaging protocol is summarized in Figure 4.
  The following imaging parameters will be acquired:
  * Biventricular end-diastolic and end-systolic volume, ejection fraction, stroke volume
  * Biventricular mass, wall thickness
  * T1 mapping; native and > 10 minutes post contrast injection as an estimate of left ventricular diffuse fibrosis and extracellular volume
  * Late enhancement for detection of regional fibrosis and scar
  * Myocardial feature tracking for analysis of deformation/motion
  * Epicardial fat volume
Diagnostic Test: Cardiopulmonary exercise testing — After completion of a regular cardiac rehabilitation program patients are scheduled to undergo their discharge examination at 3 to 4 weeks after the operation in order to be functionally characterized. Cardiopulmonary exercise testing will be performed, if possible by patients condition, on a mechanically braked bicycle ergometer and respiratory gas exchange analysis via a mouthpiece or facemask.

SUMMARY:
To evaluate the role of adipose tissue inflammation in patients with heart failure with preserved ejection fraction (HFpEF). Patients undergoing coronary artery bypass grafting with HFpEF and without heart failure will be included in this prospective study. Epicardial, paracardial, paraaortic/paravascular, subcutaneous adipose tissue samples as well as myocardial tissue will be harvested during cardiac surgery. Inflammatory patterns of these tissues and their relation to circulating markers will be investigated.

DETAILED DESCRIPTION:
Heart Failure with preserved Ejection Fraction (HFpEF) is a growing public health concern with an increasing incidence, high morbidity and mortality and no proven therapy to date. Better characterization of individual pathophysiological implications is mandatory to develop effective therapeutic strategies or preventive programs. Obesity is an important risk factor for the development of HFpEF and also modulates its course possibly by its association with systemic inflammation. However, the role of adipose tissue (AT) inflammation in the development, maintenance and functional impairments in HFpEF has been under-investigated. Dysfunctional AT leads to a shift from a protective adipokine profile to an imbalanced production of pro-inflammatory, pro-oxidant and pro-fibrotic adipokines. Besides depot specific paracrine effects, the overall secretory activity or endocrine effect of AT can be evaluated in peripheral plasma.

The investigators hypothesize that adipose inflammation distinguishes obese HFpEF patients from obese patients without heart failure and that adipose tissue inflammation is a key driver the maintenance and development of HFpEF and determines functional capacity.

In addition the investigators hypothesize that the degree of myocardial inflammatory alterations is more closely related to epicardial tissue alterations than subcutaneous or visceral AT tissue inflammation or peripheral adipokine profiles.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF: Left ventricular ejection fraction ≥ 50%, NT-pro-BNP ≥ 125ng/l, evidence of structural heart diseases (diastolic dysfunction, left ventricular-hypertrophy or left atrial-dilatation), BMI ≥ 30kg/m²
* Non-HF patients: No history of heart failure, Left ventricular ejection fraction > 50% and NT-pro-BNP <125ng/l

Exclusion Criteria:

* Previous cardiac surgery / coronary intervention / myocardial infraction
* Acute coronary syndrome (Serum levels of troponin T >50 pg/ml)
* Left ventricular ejection fraction < 50%
* Indication for concomitant valvular surgery
* Planned beating heart coronary bypass surgery
* Hemodynamic instability
* Contraindication for magnetic resonance imaging
* Pregnancy
* Age < 18 years
* No informed consent possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable patients with indication for coronary bypass crafting will be prospectively identified at the Heart Center Leipzig (either during the admission process for patients referred to surgery or at the time of coronary angiography when the indication for operative revascularization is established). Patients will be grouped according to the presence of HFpEF and obesity in order to generate 3 distinct patient groups, defined as:
  1. Obesity HFpEF
  2. Obesity Non-HF
  3. Non-Obesity Non-HF
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue inflammation | Tissue collection during surgery.
  Adipose tissue inflammation and distribution as well as association with adipokines

SECONDARY OUTCOMES:
Evaluation of serum adipokine levels | At baseline, before surgery.
  Circulating adipokine levels will be measured at a central lab.
Cardiac MRI - Myocardial function | At baseline, before surgery.
  Myocardial function and extent of myocardial fibrosis.
Cardiac MRI - Epicardial fat | At baseline, before surgery.
  Extent of epicardial fat.
Echocardiography | At baseline, before surgery and at follow-up approximately three months after surgery.
  Measurement of standard echocardiographic parameters of left- and right- ventricular systolic and diastolic function.
Functional capacity on spiroergometry | At follow-up approximately three months after surgery.
  Follow-up investigation by spiroergometry to assess post-surgical functional capacity. Measures included Peak Oxygen consumption (VO2 max) and oxygen consumption at anaerobic threshold (AT VO2)
Stress echocardiography | At follow-up approximately three months after surgery.
  Assessment of echocardiographic parameters of left- and right- ventricular systolic and diastolic function during semi-supine bicycle exercise. These measures include the change of E/E' during exercise for the left ventricle and the change of tricuspid annular plane systolic excursion (TAPSE) during exercise for the right ventricle.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Centre at University Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided